CLINICAL TRIAL: NCT06832007
Title: The Effect of Light Intervention on Recovery in Individuals With Opioid Use Disorder (OUD)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Rui Zhang, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-300014352; 31322 (Other Grant/Funding Number: BBRF)
Record Dates: First submitted 2025-02-06; First posted 2025-02-18 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Opioid Use Disorder; Sleep; Circadian Rhythms; fMRI Research
Keywords: opioid use disorder; sleep; circadian rhythms; fMRI research
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental light (Experimental): MOUD participants
  Interventions: Device: AYO light glasses (experimental)
- Comparison light (Active Comparator): MOUD participants
  Interventions: Device: AYO light glasses (comparator)
- Healthy control (No Intervention)

INTERVENTIONS:
Device: AYO light glasses (experimental) — OUD patients are asked to wear AYO light therapy glasses (wavelength 470nm ± 2nm, irradiance 250 μW/cm2 or approx.1500 m-EDI) daily for 30 min after habitual wake-up times for two weeks.
  Arms: Experimental light
Device: AYO light glasses (comparator) — The comparison group will wear the same AYO glasses but with lower intensity (1% light intensity) compared to the experimental group. This group will also self-administer 30 min of light from commercially available light glasses each morning for two weeks
  Arms: Comparison light

SUMMARY:
Opioid use disorder (OUD) is a chronic relapsing disorder and is well-known for its high-risk rate of overdoses and death. In OUD, sleep and circadian disruptions are highly prevalent, interfere with opioid maintenance treatment outcomes and increase the risk of relapse. So far, commonly used pharmacological sleep treatments fail to improve sleep or decrease illicit drug use in OUD. Thus, there is an urgent need to fill this research gap.

Previous work showed that OUD patients who were receiving opioid agonist treatment (MOUD+) exhibited greater irregularity of sleep-wake cycle. In OUD patients, sleep-wake irregularity was associated with years of heroin use and low light exposure. Bright light therapy (BLT) is a very promising circadian/sleep intervention for several sleep, psychiatric and neurological disorders. BLT improved circadian, sleep outcomes and negative mood. In a pilot study, BLT improved objective and subjective sleep in patients with alcohol use disorder. Here investigators proposed an intervention study for MOUD+ patients to determine effects of BLT as an adjunct treatment on sleep and circadian outcomes including endogenous circadian rhythm, rest-activity rhythm and sleep neurophysiology (Primary objectives); and to determine effects of BLT on brain function and on clinical outcomes including negative affect, craving and illicit drug use and whether changes in sleep and circadian rhythm mediate the BLT effect on brain recovery and clinical outcomes (Secondary objectives).

Fifty MOUD+ will be assigned either to bright light or to dim light group for 2 weeks. The groups will be matched for age, sex, race and OUD medication (Methadone vs Buprenorphine). The study will run throughout the year such that it occurs during all seasons. Light exposure will be measured with light sensor for additional control. All MOUD+ participants will have a daily 30-min light exposure (bright or dim blue light) in the morning after their habitual wake-up time and will be asked to avoid evening light before bed. Dim light melatonin onset, accelerometer, sleep EEG and questionnaires will be used to measure objective and subjective sleep and circadian outcomes. For brain function, cue-reactivity task will be used to assess brain activation during drug craving. Resting state functional connectivity and brain state dynamics will be assessed by rsfMRI. Mood, opiate craving and illicit drug use will be assessed. All measures will be repeated before and after the treatment. Investigators expect that BLT would normalize sleep and circadian outcomes, attenuate impairments in brain functions and result in better clinical outcomes. If successful, light therapy will provide add-on benefits to opioid agonist therapy and facilitate OUD recovery process.

ELIGIBILITY:
Inclusion Criteria:

* All Participants
* Between 18 and 60 years old
* Fluent in English
* Able to provide written informed consent

OUD

* DSM-5 diagnosis of an OUD.
* ≥12 months of lifetime opioid use
* Positive on urine drug screen for buprenorphine or methadone
* Receiving opioid agonist therapy for OUD (e.g., methadone or buprenorphine) with a stable dose for the past month. Must have been stabilized on OMT medication, since the increasing of doses during induction phase might interfere with outcomes and unstable patients might experience strong withdrawal symptoms in the morning which makes them unsuitable for a home-based BLT.
* Other substance use was not exclusionary, but opioids were identified as primary.

Exclusion Criteria:

All Participants

* Head trauma with loss of consciousness for more than 30 minutes as determined by medical history.
* history of seizures/epilepsy.
* Pregnant and/or currently breast-feeding.
* Presence of ferromagnetic objects in the body that are contraindicated for MRI or fear of enclosed spaces.
* Eye disease including disease of the anterior and posterior segment of the eye, cataracts, retinopathy, glaucoma, amblyopia, scotoma, color or night blindness, corneal pathologies, macular degeneration, or retinitis pigmentosa reported by history or identified by eye exam
* History of eye surgery
* Chronic migraine triggered by bright light
* worked night shift or traveled across>2 time zones in the past month

OUD

* diagnosis of substance use disorder other than for opioids that was deemed to be primary
* lifetime diagnosis of schizophrenia, bipolar disorder, or suicidality.
* History of light treatment
* Unstable dose of psychiatric medication (hypnotics, sleep aids, and antidepressants must be stable for 30 days before and during the study)

HC

* Current or past DSM-IV or DSM-5 diagnosis of a psychiatric disorder including substance use disorder (except for nicotine/caffeine).
* Current DSM-5 sleep-wake disorders including insomnia disorder

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-09-06 (Actual); Primary Completion 2028-09-16 (Estimated); Study Completion 2028-09-16 (Estimated)

PRIMARY OUTCOMES:
Dim light melatonin onset (DLMO) | the day directly before and after the intervention
  DLMO is assessed for endogenous circadian phase.Participants will be asked to remain awake in dim light < 5 lux. Salivary melatonin sample will be collected hourly and start 5h before habitual bedtime. Melatonin concentration will be later radioimmunoassayed. DLMO will be calculated as the time when melatonin concentration exceeds and remains above 4 pg/mL.
melatonin metabolites level | the day directly before and after the intervention
  Participants will be asked to collect their first morning urine void (overnight urine) upon waking. Urinary metabolite of melatonin 6-sulphatoxymelatonin (aMT6s) will be quantified and normalized to urinary creatinine concentrations to account for variations in urine concentration.
Sleep-wake regularity | From the enrollment to the end of the treatment at 24 days
  To record rest-activity/sleep-wake patterns, participants are asked to wear a triaxial accelerometer placed on the non-dominant wrist continuously throughout the study.
Total sleep duration | From the enrollment to the end of the treatment at 24 days; 2-3 nights per week
  total sleep duration (hours) will be measured by sleep EEG. Participants will be asked to wear a wireless sleep monitor device during sleep in their home environment.
N3 sleep | From the enrollment to the end of the treatment at 24 days; 2-3 nights per week
  N3 sleep (hours) will be measured by sleep EEG. Participants will be asked to wear a wireless sleep monitor device during sleep in their home environment.
REM sleep | From the enrollment to the end of the treatment at 24 days; 2-3 nights per week
  REM sleep (hours) will be measured by sleep EEG. Participants will be asked to wear a wireless sleep monitor device during sleep in their home environment.
sleep spindle | From the enrollment to the end of the treatment at 24 days; 2-3 nights per week
  Amount of sleep spindle will be measured by sleep EEG. Participants will be asked to wear a wireless sleep monitor device during sleep in their home environment.

SECONDARY OUTCOMES:
brain signiture of craving measured by cue reactivity task | the day prior to the intervention and the day after the intervention
  Participants will passively view neutral, food and opioid related pictures. Brain activity during the picture viewing will be captured.
brain functions during resting state | the day before and after light intervention
  resting state fMRI data will be collected over an 8-min period of time. Brain functional connectivity and brain state transitions will be calculated
Ecological momentary assessment (EMA) | From the enrollment to the end of the treatment at 24 days
  self-reported mood, opioid craving, withdrawal symptoms and illicit drug use will be captured by EMA surveys. The MetricWire platform will be utilized for EMA surveys. Sleep-related questions will be prompted within 1 hour of the participant's habitual wake-up time. For the OUD group, additional questions will include prior day's illicit drug use and the usage of buprenorphine and methadone (time and dose). Light therapy-related questions, including onset and offset times, adverse effects, and changes in positive and negative mood after the daily therapy session, will be collected before 1 pm. Questions on mood, craving, and pain severity will be delivered at six semi-random timepoints each day during the participant's waking hours.

OTHER OUTCOMES:
post-illumination pupil response | study visit prior to the treatment
  Upon arrival, the non-dominate eye will be dilated with Tropicamide 0.5% and Phenylephrine 2.5%. Participants are then seated in a dimly lit room (< 5 lux, background light) for 30 min to dark adapt and to ensure complete pupil dilation prior to the study. The PIPR is measured in eight, 71-second test periods in which the stimulus, either Blue (470 nm) or Red (623 nm), is presented to the dilated eye while the pupil response of the un-dilated eye is measured (consensual pupil response). During a test period, after an initial 20-second fixation period, the stimulus is presented for 1 second followed by a 50-second recording period. The red stimulus primarily serves as a control for any nonspecific influences on the PIPR.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States